CLINICAL TRIAL: NCT05600192
Title: Target Mitochondrial Fitness, Chronobiology and Metabolism
Acronym: PI19/00507
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI19/00507
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects
Keywords: Mitochondrial fitness; Metabolism; Chronobiology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise arm (Experimental): Subjects perfom aerobic or anaerobic exercise in the morning or in the afternoon
  Interventions: Other: Aerobic or anaerobic exercise

INTERVENTIONS:
Other: Aerobic or anaerobic exercise — Aerobic or anaerobic exercise in the morning or in the afternoon

SUMMARY:
Exercise could be an element that affects the biochemical, metabolic and microbiome parameters of organisms. Thus, to identify and validate the effects of aerobic and anaerobic exercises at different times of the day (morning or afternoon) on mitochondrial fitness and whether this changes could have a relation with metabolism and cardiovascular parameters and microbiome is of great interest for its applicability in biomedicine.

As specific objectives of this project will study:

1. - To study the direct effect of aerobic and anaerobic exercise at different time points in the day on mitochondria fitness (short study: basal, at the end of the exercise and 2 h after exercise).
2. - To study mitochondria fitness under morning or afternoon aerobic and anaerobic exercise (prospective study: basal, 4, 8 and 12 weeks of the study).
3. - To identify and validate modulators and target proteins of mitochondria fitness affected by exercise (miRNA omic and proteomic analysis of mitochondria from the different groups of the study at basal and 12 weeks of the study).
4. - To study the relationship of the mitochondrial response (Objectives 1 and 2) to the different combination of exercises and chronobiology with anthropometric-clinical, carbohydrate and lipid metabolic and cardiovascular changes.
5. - To check the effect of morning or afternoon aerobic and anaerobic exercise on gut microbiota and its relation to mitochondria fitness, clinical and metabolic parameters (basal, 4, 8 and 12 weeks of the study).

ELIGIBILITY:
Inclusion Criteria:

* 20-
* IMC <30 kg/m2
* Informed consent

Exclusion Criteria:

* Smoker
* Previous physical exercise of more than 20 minutes / 2 times a week

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | From baseline to week 12
  Weight in kg
BMI (body mass index) changes | From baseline to week 12
  Measured by body composition analysis
Change in waist circumference | From baseline to week 12
  Circumference in cm
Change in hip circumference | From baseline to week 12
  Circumference in cm
Changes in diastolic and systolic blood pressure | From baseline to week 12
  To analyze the effect of exercise on blood pressure
Changes in body composition | From baseline to week 12
  To analyze the effect of exercise on anthropometric parameters measured by bioelectrical impedance analysis
Change in glucose concentration | From baseline to week 12
  Glucose in mg/dl
Change in insulin concentration | From baseline to week 12
  Insulin in mg/dl
Change in glycated haemoglobin concentration | From baseline to week 12
  Glycated haemoglobin in mg/dl
Change in Triglycerides concentration | From baseline to week 12
  Triglycerides in mg/dl
Change in cholesterol concentration | From baseline to week 12
  Serum cholesterol in mg/dl
Change in HDL concentration | From baseline to week 12
  Serum HDL in mg/dl
Change in LDL concentration | From baseline to week 12
  Serum LDL in mg/dl
Change in transaminases concentration | From baseline to week 12
  Serum transaminases in UI/l
Change in creatinine concentration | From baseline to week 12
  Creatinine in mg/dl
Change in uric acid concentration | From baseline to week 12
  Uric acid in mg/dl
Change in alkaline phosphatase concentration | From baseline to week 12
  Serum alkaline phosphatase in UI/l
Change in bilirubin concentration | From baseline to week 12
  Serum bilirubin in mg/dl
Change in lactate concentration | From baseline to week 12
  Serum lactate in mmol/L
Change in cortisol concentration | From baseline to week 12
  Serum cortisol in nmol/L
Change in total and free testosterone concentration | From baseline to week 12
  Serum total and free testosterone in nmol/L
Change in melatonine concentration | From baseline to week 12
  Serum melatonine in pg/ml
Characterize exercise participant behavior | From baseline to week 12
  International Physical Activity Questionnaire (IPAQ). The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) carried out in the last seven days, as well as walking and sitting time in a work day. It evaluates three characteristics of physics (PA): intensity (mild, moderate or vigorous), frequency (days per week) and duration (time per day). Weekly activity is recorded in Mets (Metabolic Equivalent of Task or Metabolic Index Units) per minute and week.
Mediterranean diet adherence questionnaire | From baseline to week 12
  To evaluate adherence to a Mediterranean diet pattern. It consists of 14 items in which different components of the Mediterranean diet are evaluated (number of pieces of fruit consumed per day, number of portions of legumes consumed per week...). Each item is scored as 0 or 1. A total score of <9 indicates poor adherence, while a score of ≥9 indicates good adherence.
Change in faecal microbiota | From baseline to week 12
  To evaluate faecal microbiota composition in the studied subjects and the effect of aerobic and anaerobic exercise in the morning or afternoon on faecal microbiota composition. 16S rRNA amplicons of fecal community DNA
Change in fitness mitochondrial | From baseline to week 12
  To evaluate the effect of aerobic and anaerobic exercise in the morning or afternoon on mitochondrial fitness, evaluated by mitochondrial gene expression and protein abundance, mitochondrial metabolites, mitochondrial markers trough flow citometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mora Murri Pierri, PhD, Principal Investigator — Hospital Universitario Virgen de la Victoria
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain